CLINICAL TRIAL: NCT04814966
Title: Prospective Observational Study on the Use of Extended Haemodynamic Monitoring in the Post-Anesthesia Care Unit (PACU) Using Non-invasive Methods: Feasibility and Influence on Volume Therapy and Catecholamine Treatment.
Brief Title: Feasibility of Extended Non-invasive Haemodynamic Monitoring in the PACU
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Clinical Professor, University Hospital Schleswig-Holstein
Other Study IDs: IN-PACU-02
Record Dates: First submitted 2019-07-16; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Goal Directed Therapy; Postoperative Complications; Complications; Ultrasound Therapy
Keywords: Goal directed haemodynamic optimization; Ultrasound Therapy; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-operative monitoring of all patients after anaesthesia in the post anaesthesia care unit (PACU) is standard of care today. It helps to reduce morbidity and even mortality in high-risk patients.

In addition to clinical monitoring by qualified personnel, this monitoring also includes, commonly non-invasive, intermittent, haemodynamic monitoring. This monitoring is also used to evaluate the transferability of patients from the PACU to the ward.

The aim of our study is to perform extended monitoring of volume status and haemodynamics with non-invasive monitoring methods such as transthoracic echocardiography and the volume clamp method in the recovery room.

DETAILED DESCRIPTION:
Postoperative haemodynamic management, with particular emphasis on adequate volume status, is essential for patient outcome, as is optimised intraoperative management. Postoperative monitoring is usually performed in the PACU by non-invasive, continuous and intermittent monitoring. ECG and oxygen saturation are monitored continuously, blood pressure and laboratory analyses intermittently. The assessment of adequate oxygen supply (cardiac output - haemoglobin concentration - oxygen saturation) in the PACU is traditionally approximated only by surrogate parameters such as blood pressure and heart rate, in the sense of an empirical approach. The aim should be to transfer the available data on the benefit of early, goal-oriented haemodynamic optimisation by means of extended haemodynamic monitoring to the sensitive area of the PACU. An important prerequisite for the implementation of such haemodynamic optimisation protocols is the use of non-invasive monitoring methods, which ideally provide continuous flow and pressure-based parameters in combination with the use of intermittent transthoracic echocardiography. The necessity to continue extended haemodynamic monitoring in selected patients in the PACU on the basis of non-invasive procedures is under discussion and is not part of a defined standard today (Gruenewald et al. Anaesthesia 2015). A number of non-invasive haemodynamic monitoring methods have become available over the last few years, with a large number of scientific evaluation studies investigating the methods in various clinical settings in comparison to invasive systems. Of interest for routine clinical use are the so-called volume clamp procedures, which allow non-invasive, continuous recording of haemodynamic parameters such as stroke volume, cardiac output, blood pressure and plus pressure variation. Thus, in combination with oxygen saturation and intermittent haemoglobin determinations, they enable a punctual determination of oxygen supply (Meidert et al. Front Med (Lausanne) 2017 and Renner et al. Br J Anaesth 2017).

It is of interest whether the volume clamp method in particular provides the aforementioned parameters such as blood pressure, stroke volume, cardiac output and the pulse pressure variation continuously and without interference in the awake patient in the PACU. Another aspect is the assessment of the volume status and cardiac performance that patients show on admission to the PACU. Here, special attention is paid to the volume status after the patients have been haemodynamically optimised intraoperatively with an invasive procedure. Furthermore, we will compare how the cardiac output determined by echocardiography on admission differs from the cardiac output of the volume clamp method on admission. The differences between invasive blood pressure measurement and non-invasive pressure measurement will also be assessed.

In addition, the investigators analyse the frequencies of decreased blood pressures in comparison to a patient collective that was monitored according to standard-of-care in the PACU. Also, the comparative observation of the number of interventions performed, such as volume administration and/or catecholamine administration, between the groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with ASA classification I-III undergoing abdominal surgery, surgery in urology or vascular surgery
* written consent

Exclusion Criteria:

* Age <18 years
* ASA classification IV or higher
* legal care relationship
* missing or faulty written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ASA classification I-III undergoing abdominal surgery, surgery in urology or vascular surgery and delivered to postanaesthesia care unit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
length of stay in the recovery room | up to 24 weeks
  evaluated using the Whites-Fast-Trac Scoring System
acute renal failure | up to 24 weeks
  number of short-term postoperative complications
pericardial effusion | up to 24 weeks
  number of short-term postoperative complications
pulmonary oedema | up to 24 weeks
  number of short-term postoperative complications

SECONDARY OUTCOMES:
cardiac output by echocardiography | up to 24 weeks
  cardiac output determined by echocardiography on admission
cardiac output volume clamp method | up to 24 weeks
  cardiac output determined by volume clamp method on admission
frequencies of decreased blood pressure values | up to 24 weeks
  frequencies of decreased blood pressure values between the groups
number of interventions | up to 24 weeks
  comparative observation of the number of interventions performed between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Deutschland (deu), Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldrete JA, Kroulik D. A postanesthetic recovery score. Anesth Analg. 1970 Nov-Dec;49(6):924-34. No abstract available. PMID 5534693
- [Background] Truong L, Moran JL, Blum P. Post anaesthesia care unit discharge: a clinical scoring system versus traditional time-based criteria. Anaesth Intensive Care. 2004 Feb;32(1):33-42. doi: 10.1177/0310057X0403200106. PMID 15058119
- [Background] McLaren JM, Reynolds JA, Cox MM, Lyall JS, McCarthy M, McNoble EM, Petersen VR. Decreasing the length of stay in phase I postanesthesia care unit: an evidence-based approach. J Perianesth Nurs. 2015 Apr;30(2):116-23. doi: 10.1016/j.jopan.2014.05.010. PMID 25813297
- [Background] Jain A, Muralidhar V, Aneja S, Sharma AK. A prospective observational study comparing criteria-based discharge method with traditional time-based discharge method for discharging patients from post-anaesthesia care unit undergoing ambulatory or outpatient minor surgeries under general anaesthesia. Indian J Anaesth. 2018 Jan;62(1):61-65. doi: 10.4103/ija.IJA_549_17. PMID 29416152
- [Background] Eichenberger AS, Haller G, Cheseaux N, Lechappe V, Garnerin P, Walder B. A clinical pathway in a post-anaesthesia care unit to reduce length of stay, mortality and unplanned intensive care unit admission. Eur J Anaesthesiol. 2011 Dec;28(12):859-66. doi: 10.1097/EJA.0b013e328347dff5. PMID 21885983
- [Background] Waddle JP, Evers AS, Piccirillo JF. Postanesthesia care unit length of stay: quantifying and assessing dependent factors. Anesth Analg. 1998 Sep;87(3):628-33. doi: 10.1097/00000539-199809000-00026. PMID 9728843
- [Background] Samad K, Khan M, Hameedullah, Khan FA, Hamid M, Khan FH. Unplanned prolonged postanaesthesia care unit length of stay and factors affecting it. J Pak Med Assoc. 2006 Mar;56(3):108-12. PMID 16696508
- [Background] Ameloot K, Van De Vijver K, Van Regenmortel N, De Laet I, Schoonheydt K, Dits H, Broch O, Bein B, Malbrain ML. Validation study of Nexfin(R) continuous non-invasive blood pressure monitoring in critically ill adult patients. Minerva Anestesiol. 2014 Dec;80(12):1294-301. Epub 2014 Apr 4. PMID 24705004
- [Background] Batz G, Dinkel M. [Hemodynamic monitoring - imaging procedures / cardiac ultrasound]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2016 Oct;51(10):626-634. doi: 10.1055/s-0041-110009. Epub 2016 Oct 20. German. PMID 27764871
- [Background] Broch O, Renner J, Gruenewald M, Meybohm P, Schottler J, Caliebe A, Steinfath M, Malbrain M, Bein B. A comparison of the Nexfin(R) and transcardiopulmonary thermodilution to estimate cardiac output during coronary artery surgery. Anaesthesia. 2012 Apr;67(4):377-83. doi: 10.1111/j.1365-2044.2011.07018.x. Epub 2012 Feb 11. PMID 22324797
- [Background] Pouwels S, Lascaris B, Nienhuijs SW, Arthur Bouwman R, Buise MP. Validation of the Nexfin(R) non-invasive continuous blood pressure monitoring validated against Riva-Rocci/Korotkoff in a bariatric patient population. J Clin Anesth. 2017 Jun;39:89-95. doi: 10.1016/j.jclinane.2017.03.029. Epub 2017 Mar 31. PMID 28494917
- [Background] White PF, Song D. New criteria for fast-tracking after outpatient anesthesia: a comparison with the modified Aldrete's scoring system. Anesth Analg. 1999 May;88(5):1069-72. doi: 10.1097/00000539-199905000-00018. No abstract available. PMID 10320170
- [Background] Broch O, Carstens A, Gruenewald M, Nischelsky E, Vellmer L, Bein B, Aselmann H, Steinfath M, Renner J. Non-invasive hemodynamic optimization in major abdominal surgery: a feasibility study. Minerva Anestesiol. 2016 Nov;82(11):1158-1169. Epub 2016 Jun 28. PMID 27352070
- [Background] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849
- [Background] Gruenewald M, Renner J. Do we need to monitor cardiac output in spontaneously breathing patients? Anaesthesia. 2015 Feb;70(2):122-5. doi: 10.1111/anae.12951. No abstract available. PMID 25583187
- [Background] Meidert AS, Saugel B. Techniques for Non-Invasive Monitoring of Arterial Blood Pressure. Front Med (Lausanne). 2018 Jan 8;4:231. doi: 10.3389/fmed.2017.00231. eCollection 2017. PMID 29359130
- [Background] Renner J, Gruenewald M, Hill M, Mangelsdorff L, Aselmann H, Ilies C, Steinfath M, Broch O. Non-invasive assessment of fluid responsiveness using CNAP technology is interchangeable with invasive arterial measurements during major open abdominal surgery. Br J Anaesth. 2017 Jan;118(1):58-67. doi: 10.1093/bja/aew399. PMID 28039242